CLINICAL TRIAL: NCT01510964
Title: The Involvement of Breast Cancer Patients During Oncological Consultations. A Multi-centre Randomized Controlled Trial. The Study Protocol
Brief Title: The Involvement of Breast Cancer Patients During Oncological Consultations
Acronym: INCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: INCA (CE.Prot. 1719)
Record Dates: First submitted 2011-12-22; First posted 2012-01-18 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2011-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Patient involvement; Question prompt-sheet; Doctor-patient communication; RCT
MeSH Terms: conditions — Breast Neoplasms; Patient Participation | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- prompt-sheet (Experimental): Patients and companions of intervention group receive a form on which to write their reply to the following request: "Please indicate the arguments which you want to discuss today with your oncologist" and the prompt sheet. An introduction explains the importance of asking questions during the consultations. The patient (companion) is invited to select among a written list of about 50 possible questions those, if any, s/he would like to ask today to the oncology.
  Interventions: Behavioral: prompt-sheet
- control group (Other): Patients and companions of the control group receive a form on which to write their reply to the following request: "Please indicate the arguments which you want to discuss today with your oncologist"
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: prompt-sheet — Prompt sheet is a form on which to write the reply to the following request: "Please indicate the arguments which you want to discuss today with your oncologist" and a written list of possible questions the patient (companion) would like to ask to the oncology.
  Arms: prompt-sheet
Behavioral: control group — Patients and companions of the control group receive a form on which to write their reply to the following request: "Please indicate the arguments which you want to discuss today with your oncologist"
  Arms: control group

SUMMARY:
The main aim of the study is to assess if a pre consultation intervention facilitates greater participation of patients (and accompanying key persons when present) in the consultation process by determining an increase in questioning and/or in the number of different illness related issues (e.g. diagnosis, treatment, prognosis) being discussed with the oncologist.

Other aims are to assess the effect of the intervention on the oncologist's level of patient involvement, on patient satisfaction and coping and to explore the role of key persons accompanying the patient.

The investigators expect that patients who have the opportunity to rehearse their informative needs before the consultation will ask a greater number of questions which in turn will determine their greater involvement by the physician and a greater number of satisfied needs. The investigators expect also that the straightforward use of a list of printed questions of potential relevance for cancer patients and their companions at an early stage of illness, by modifying the process of information exchange, increases their participation and satisfaction with the consultation, with potential benefits for treatment adherence and consequently treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients
* age between 18 and 75 years
* attending the Oncology Out-patient Clinics of the participating centres
* recent diagnosis of breast cancer at an early stage

Exclusion Criteria:

* presence of metastasis or relapse
* severe mental deterioration
* comprehension difficulties of the Italian language.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
number of question during the consultation | 1 hour after the intervention (question prompt-sheet)
  The intervention prompt-sheet aims to increase the number of question by giving the opportunity to patients and companions to reflect on their informative needs on the basis of a wide range of possible questions from which to choose those perceived as most relevant in view of the subsequent consultation. Question asking is considered an index for patient participation during the consultation. The total number of patient questions during the consultation regarding diagnosis, prognosis, treatment and other issues is the primary outcome measure.

SECONDARY OUTCOMES:
The number of informative needs not met during the consultation. | 1 hour after the intervention (question prompt-sheet)
  This measure is derived by comparing the number of questions indicated by patients and their companion before the consultation with those actually raised during the consultation
Ability to cope with the illness | 2 hours after the intervention (question prompt-sheet)
  the Patient Enablement Instrument (PEI) is a questionnaire of six items on a Likert scale from 0 (same or less) to 2 (much better, much more), administered after the consultation.
Patient involvement (SDM-Q and OPTION) | 2 hours after the intervention (question prompt-sheet)
  The SDM-Q is a self administered questionnaire of 9 items on a Likert scale from 1 to 6 and assesses patients' perception of the decisional process and their level of involvement during the consultation. The OPTION Scale is composed of 12 items of operational definitions of different patient involving skills, rated on a Likert scale from 0 to 4. The scale is applied by trained raters to the audio-recording of the consultation
Satisfaction with decisions (SWD). | 2 hours after the intervention (question prompt-sheet)
  Satisfaction with Decision Scale (SWD) is a questionnaireof 6 items on a Likert scale from 0 (completely disagree) to 5 (agree completely), administered after the consultation.
Recalling and understanding of information | 2 hours after the intervention (question prompt-sheet)
  The Recall Questionnaire consists of six questions which ask the patient's to recall the received information on treatment decisions and pathology. We added three other questions, rated on a 0 (no at al) to 5 (very much) likert scale asking whether the patient succeeded in their purpose of question asking, whether the oncologist answered the questions properly and how much more information she would have needed.
Overall consultation atmosphere (VR-COPE, RIAS, AIMIT on the audio-recorded consultation) | 1 hour after the intervention (question prompt-sheet)
  VRCOPE assesses the content, the process and relational aspects of patient-centred communication during medical consultations on the basis of a multidimensional evaluation and comprises nine items. RIAS is a coding system of medical consultations, composed by 40 categories describing interactions between doctors and patients. AIMIT is a coding system to assess in the therapeutic dialogue the activity of interpersonal motivational systems that guide the verbal and non verbal behaviors during interactions.
Perceived Patient-doctor relationship (PDRQ-9 and DDPRQ-10) | 2 hours after the intervention (question prompt-sheet)
  PDRQ-9 is a self-administered (after the consultation) questionnaire of 9 items on a Likert scale from 1 to 5, to measure the relationship between the doctor and the patient, from a patient point of view.The DDPRQ-10 is a self-report instrument of 10 items on a Likert scale from 1 to 6, completed by physicians after an encounter with a patient.
Perceived role preference of the patient (CPS) | 2 hours after the intervention (question prompt-sheet)
  CPS (Oncologist version) assesses how the oncologist perceives the role that patient might prefer regarding the decision making process.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Goss, Principal Investigator — Universita di Verona
Locations (1):
- Azienda Ospedaliera Universitaria Integrata, Verona, Italy

REFERENCES:
- [Derived] Buizza C, Cela H, Ferrari C, Goss C, Bottacini A, Mazzi MA, Del Piccolo L, Ghilardi A. Does being accompanied make a difference in communication during breast cancer consultations? Results from a multi-centered randomized controlled trial. J Psychosoc Oncol. 2021;39(2):189-203. doi: 10.1080/07347332.2020.1829775. Epub 2020 Oct 22. PMID 33089767
- [Derived] Buizza C, Ghilardi A, Mazzardi P, Barbera D, Fremondi V, Bottacini A, Mazzi MA, Goss C. Effects of a Question Prompt Sheet on the Oncologist-Patient Relationship: a Multi-centred Randomised Controlled Trial in Breast Cancer. J Cancer Educ. 2020 Jun;35(3):621-628. doi: 10.1007/s13187-019-01505-6. PMID 30852786
- [Derived] Bottacini A, Goss C, Mazzi MA, Ghilardi A, Buizza C, Molino A, Fiorio E, Nortilli R, Amoroso V, Vassalli L, Brown RF. The involvement of early stage breast cancer patients during oncology consultations in Italy: a multi-centred, randomized controlled trial of a question prompt sheet versus question listing. BMJ Open. 2017 Aug 11;7(8):e015079. doi: 10.1136/bmjopen-2016-015079. PMID 28801395
- [Derived] Goss C, Ghilardi A, Deledda G, Buizza C, Bottacini A, Del Piccolo L, Rimondini M, Chiodera F, Mazzi MA, Ballarin M, Bighelli I, Strepparava MG, Molino A, Fiorio E, Nortilli R, Caliolo C, Zuliani S, Auriemma A, Maspero F, Simoncini EL, Ragni F, Brown R, Zimmermann C. INvolvement of breast CAncer patients during oncological consultations: a multicentre randomised controlled trial--the INCA study protocol. BMJ Open. 2013 May 2;3(5):e002266. doi: 10.1136/bmjopen-2012-002266. PMID 23645911